CLINICAL TRIAL: NCT01933451
Title: Postoperative Lung Function, Kidney Function, Inflammatory Response and Short-term Outcome After Esophagectomy and Reconstruction: Intraoperative Fluid Management Controlled With Lower and Higher Pulse Pressure Variation
Brief Title: Outcome Study of Restrictive vs. Liberal Intraoperative Fluid Management Guided by PPV in Esophagectomy
Acronym: PPV
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The grant for this study was not allowed.
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 201211078RIB
Record Dates: First submitted 2013-03-19; First posted 2013-09-02 (Estimated); Last update posted 2013-09-02 (Estimated); Status verified 2013-03

CONDITIONS: Other Complications of Esophagostomy
Keywords: fluid therapy; Intraoperative care; Patient Outcome Assessment; pulse pressure variation; restrictive fluid therapy; goal-directed fluid therapy; esophagectomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Restrictive intraoperative fluid therapy (Experimental): To Keep intraoperative pulse pressure variation above 18%.
  Interventions: Other: Intraoperative fluid therapy
- Liberal intraoperative fluid therapy (Other): To keep intraoperative pulse pressure variation below 13%.
  Interventions: Other: Intraoperative fluid therapy

INTERVENTIONS:
Other: Intraoperative fluid therapy — Intraoperative fluid therapy is directed by pulse pressure variation to a setting value, above 18% or below 13%.

SUMMARY:
The purpose of this study is to determine whether intraoperative restrictive fluid management guided by pulse pressure variation produces a better effect on the postoperative lung function, kidney function, inflammatory response and short-term outcome after esophagectomy and reconstruction.

DETAILED DESCRIPTION:
Measurements: intraoperative Lung injury score, Lung water index, Pulmonary vascular Permeability Index Measurements: intraoperative and postoperative Plasma creatine, C reactive protein (CRP), lactate, Neutrophil gelatinase-associated lipocalin (NGAL), Interleukin-6 (IL-6), Interleukin-8 (IL-8)

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing esophagectomy and reconstruction

Exclusion Criteria:

* ASA score >= 3, (American Society of Anesthesiologist physical status classification system)
* arrythmia, atrial fibrillation
* lung diseases, such as COPD (chronic obstructive pulmonary disease); lung function test showed moderate to severe ventilation defect
* plasma creatinine level above 1.5 mg/dl

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-03; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
postoperative lung function, kidney function, inflammatory response | from introperative to postoperative day 2
  plasma creatinine, CRP, lactate, NGAL, IL-6, IL-8

SECONDARY OUTCOMES:
postoperative short-term outcome | the duration of hospital stay, about 4 weeks
  Respiratory complication, cardiovascular complication, acute renal failure, another complications

CONTACTS AND LOCATIONS:
Overall Officials: Ya-Uyng Cheng, MD. PHD., Principal Investigator — chengyj@ntu.edu.tw
Locations (1):
- Department of Anesthesiology, National Taiwan University Hospital, Taipei, Taiwan